CLINICAL TRIAL: NCT01900613
Title: Niños Sanos, Familia Sana (Healthy Children/Healthy Family): A Multi-Intervention Program to Prevent Childhood Obesity in Mexican-Heritage Children in Rural California
Brief Title: Niños Sanos, Familia Sana - A Multi-Intervention Program to Prevent Childhood Obesity in Mexican-Heritage Children in Rural California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 216443
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: child obesity; Mexican-American; Nutrition education; Intervention
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Niños Sanos Familia Sana consists of CBPR developed nutrition education and economic vouchers for fruit and vegetable purchase in Firebaugh supermarket
  Interventions: Behavioral: Ninos Sanos Familia Sana
- Comparison (Active Comparator): Comparison community of San Joaquin
  Interventions: Behavioral: Ninos Sanos Familia Sana

INTERVENTIONS:
Behavioral: Ninos Sanos Familia Sana

SUMMARY:
Obesity and overweight are health problems resulting from the interaction of predisposing genes with environmental, economic and social stimuli, in conjunction with excess caloric intake throughout growth from childhood to adulthood. Evidence suggests that a major barrier in controlling overweight/obesity is the complex interrelation of these factors, making single-approach interventions less likely to succeed than integrated, multi-faceted approaches. The proposed project aims to deliver a multi-faceted behavioral intervention developed over the past 18 months by a university-community /school-based collaborative. This project aims to provide new knowledge about the effectiveness of interventions designed specifically to achieve successful weight management among Mexican-origin children ages 3-8, and identify associated mediating factors. Deliverables will include community-based, collaborative and sustainable tools to support weight-management goals in this demographic. UC Davis and UC Cooperative Extension (UCCE) faculty form the investigator team, collaborating on key decision points with the project community in California's Central Valley. The investigators hypothesize that the identified mediating factors will increase fruit and vegetable consumption. The investigators also hypothesize an increase in the intensity and frequency of physical activity among children in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Family with child between ages 3-8 years

Exclusion Criteria:

* None

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Child BMI | 3 years
  Over 3 years child increases in child BMI will be decreased

SECONDARY OUTCOMES:
Parent BMI | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Adela de la Torre, PhD, Principal Investigator — Center for Transnational Health, UC Davis
Locations (1):
- UC Davis, Davis, California, United States

REFERENCES:
- [Background] Haworth CM, Dale PS, Plomin R. The etiology of science performance: decreasing heritability and increasing importance of the shared environment from 9 to 12 years of age. Child Dev. 2009 May-Jun;80(3):662-73. doi: 10.1111/j.1467-8624.2009.01289.x. PMID 19489895
- [Background] Sinha A, Kling S. A review of adolescent obesity: prevalence, etiology, and treatment. Obes Surg. 2009 Jan;19(1):113-20. doi: 10.1007/s11695-008-9650-4. Epub 2008 Aug 30. PMID 18758874
- [Background] Dobbins M, De Corby K, Robeson P, Husson H, Tirilis D. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6-18. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD007651. doi: 10.1002/14651858.CD007651. PMID 19160341
- [Derived] Sadeghi B, Kaiser LL, Hanbury MM, Tseregounis IE, Shaikh U, Gomez-Camacho R, Cheung RCY, Aguilera AL, Whent L, de la Torre A. A three-year multifaceted intervention to prevent obesity in children of Mexican-heritage. BMC Public Health. 2019 May 16;19(1):582. doi: 10.1186/s12889-019-6897-8. PMID 31096944
- [Derived] de la Torre A, Sadeghi B, Green RD, Kaiser LL, Flores YG, Jackson CF, Shaikh U, Whent L, Schaefer SE. Ninos Sanos, Familia Sana: Mexican immigrant study protocol for a multifaceted CBPR intervention to combat childhood obesity in two rural California towns. BMC Public Health. 2013 Oct 31;13:1033. doi: 10.1186/1471-2458-13-1033. PMID 24172250